CLINICAL TRIAL: NCT04394663
Title: High Dose Oral Omeprazole Versus Standard Continuous Intravenous Pantoprazole in Patient With Peptic Ulcer Bleeding and Undergo Successful Therapeutic Endoscopy; Non-inferiority Randomized Controlled Trial
Brief Title: High Dose Oral Omeprazole in High Risk UGIB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Principle investigator, Gastrointestinal Unit, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP019
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: GI Bleeding
Keywords: oral proton pump inhibitor
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: The patients with successful endoscopic hemostasis in peptic ulcer bleeding were equally randomized to either high-dose oral PPI or standard IV PPI for 3 days
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not know the assigned treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose oral PPI (Experimental): Omeprazole 80 mg/day (40 mg twice a day) per oral route for 72 hours
  Interventions: Drug: High-dose oral omeprazole
- Standard IV PPI (Active Comparator): Pantoprazole 8 mg/hour IV continuous drip for 72 hours
  Interventions: Drug: Standard IV PPI

INTERVENTIONS:
Drug: High-dose oral omeprazole — Local made oral omeprazole 40 mg twice daily will be prescribed for 72 hours after randomization.
  Arms: High-dose oral PPI
Drug: Standard IV PPI — Pantoprazole 8mg/hour IV continuous drip will be prescribed for 72 hours after randomization
  Arms: Standard IV PPI

SUMMARY:
Peptic ulcer bleeding is the most common etiology in upper gastrointestinal bleeding all over the world. After endoscopic treatment, proton pump inhibitor (PPI) is recommended to prevent re-bleeding. Intravenous PPI is recommended as a standard treatment. In the past, there were many trials showing the efficacy of high-dose oral PPI after endoscopic hemostasis but most were industrial sponsor which assessing an expensive PPI. Moreover, the number of patients in those studies were insufficient to confirm a non-inferiority outcome in term of rebleeding by using oral PPI. This study will evaluate a high-dose, local-made PPI (omeprazole) in peptic ulcer treatment after successful endoscopic hemostasis compared to standard IV PPI continuous drip in term of rebleeding, as well as 24-hour gastric pH monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peptic ulcer bleeding and endoscopic finding show ulcer with Forrest classification Ia (spurting haemorrhage), IIa (oozing haemorrhage), Ib (non-bleeding visible vessel)
* Age > 18 years old

Exclusion Criteria:

* Deny to participate
* Pregnancy or lactation
* Low risk peptic ulcer bleeding including clean base ulcer, flat pigmented spot
* Non-peptic ulcer bleeding eg. erosive gastritis/duodenitis, Mallory Weiss tear, esophageal/gastric/duodenal varices, vascular lesions (eg. Dieulafoy) , malignant ulcer
* Bleeding tendency
* Terminal stage of cancer
* ESRD on hemodialysis
* Decompensated liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of 3-day peptic ulcer rebleeding | 3 days

SECONDARY OUTCOMES:
Percentage of 24-hour gastric pH above 6 | 3 days
Rate of 30-day peptic ulcer rebleeding | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Rapat Pittayanon, MD, Principal Investigator — King Chulalongkorn Memorial Hospital
Locations (2):
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok
  - Surin Hospital, Surin